CLINICAL TRIAL: NCT05772195
Title: Safer Services, Organisations, and Innovation: The Central London Patient Safety Research Collaboration
Brief Title: Central London Patient Safety Research Collaboration
Status: Active, not recruiting | Type: Observational
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Charles Matthew Oliver, Associate Professor, University College London Hospitals
Other Study IDs: NIHR204297
Record Dates: First submitted 2023-01-05; First posted 2023-03-16 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Surgery-Complications; Safety Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Before major system reorganisation: Theme 1 - elective recovery plan 2017/18-2019/20
- Before major system reorganisation - intra-pandemic: Theme 1 - elective recovery plan 2020/21-2021/22
- Post system reorganisation: Theme 1 - elective recovery plan 2023/24 and 2024/25

SUMMARY:
Patient safety is a priority for healthcare systems. In safe systems, patients would be saved from avoidable harm, both from their own conditions, and from the care and treatments provided to them. Amongst the highest risk clinical settings are Surgical, Perioperative, Acute and Critical carE services (SPACE).

The Central London Patient Safety Research Collaborative is funded to deliver world-class research into improving the safety of SPACE services, within which the investigators will evaluate major service reorganisation, compare and investigate organisational safety and quality, and investigate the disparity in postoperative complications associated with socioeconomic factors.

DETAILED DESCRIPTION:
Patient safety is a priority for healthcare systems. In safe systems, patients would be saved from avoidable harm, both from their own conditions, and from the care and treatments provided to them.

International estimates suggest that of 421 million hospitalisations worldwide annually, there are 42.7 million adverse events or unsafe experiences, making avoidable harm the 14th leading cause of death and serious illness. Amongst the highest risk clinical settings are Surgical, Perioperative, Acute and Critical carE services (SPACE), treating >25 million NHS patients annually. Patient safety risks are particularly likely in these environments, both because of what clinicians are required to do (the trauma of surgery and anaesthesia, the need for rapid recognition and decision-making in acute illness) and the patient's condition (because acute illness and surgery compound the risks from long-term conditions such as diabetes and heart disease).

The Central London Patient Safety Research Collaborative will be funded by the NIHR to deliver world-class research into improving the safety of Surgical, Perioperative, Acute and Critical carE services (SPACE) services. Three themes, using existing patient data, are included in this application:

1. Safer services The investigators will evaluate the safety of SPACE-related interventions of the NHS' post-pandemic Elective Recovery Plan. The investigators will use NHS administrative datasets to identify and explore changes in safety and quality over the implementation timeframe using advanced statistical methods.
2. Safer organisations From linked clinical and administrative datasets, The investigators will identify and seek to contextualise high- and low-performing units and hospitals across SPACE services using advanced statistical methods. This work will be followed by qualitative research, exploring why differences exist.
3. Safer innovations The investigators will identify the timeframe over which patients from deprived backgrounds develop worse postoperative outcomes (as has previously been demonstrated). These novel findings could pave the way for interventions to reduce inequality.

ELIGIBILITY:
Inclusion Criteria:

* as determined by clinical audits

Exclusion Criteria:

* missing key data items/ or linkage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major surgery Critical care admission
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Total number of elective operations performed within the NHS | 8 years (2017/18 - 2024/25) as per cohort definitions
  Process and outcomes following major system change (Theme 1):
  To be presented and analysed
  1. nationally,
  2. regionally and
  3. at hospital Trust- level
  To assess the effectiveness of the NHS Elective recovery plan (https://www.england.nhs.uk/2022/02/nhs-publishes-electives-recovery-plan-to-boost-capacity-and-give-power-to-patients/)
Incidence/prevalence of postoperative complications | Pre 2023
  Process and outcomes following major system change (Theme 1):
  Postoperative complications.
  * Occurring whilst inpatient, following the index surgical procedure.
  * Classified using the Clavien-Dindo and Postoperative Morbidity Survey systems
  * We will gather and link data from national audit and registry datasets.
  * We will compare patient outcomes within and between organisations to investigate safety and quality
Incidence/prevalence of postoperative complications stratified by socioeconomic and ethnic descriptors | Pre 2023
  Theme 3 safer innovations:
  Postoperative complications.
  * Occurring whilst inpatient, following the index surgical procedure.
  * Classified using the Clavien-Dindo and Postoperative Morbidity Survey systems
  * We will gather and link data from national audit and registry datasets.
  * We will investigate divergences in patient outcomes, stratified by socioeconomic and ethnic descriptors

SECONDARY OUTCOMES:
Mean/median postoperative length of stay (days) | 8 years (2017/18 - 2024/25) as per cohort definitions
  Theme 1: Health economic assessment of the implementation of the NHS Elective recovery plan
Mean/Median postoperative critical care length of stay (days) | 8 years (2017/18 - 2024/25) as per cohort definitions
  Theme 1: Health economic assessment of the implementation of the NHS Elective recovery plan

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom